CLINICAL TRIAL: NCT06225128
Title: Dynamics of Resistance Emergence to Azacitidine-based Therapies in Acute Myeloid
Brief Title: Dynamics of Resistance Emergence to Azacitidine-based Therapies in Acute Myeloid Leukemia
Acronym: DREAM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230805
Record Dates: First submitted 2023-12-12; First posted 2024-01-25 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with AML
  Interventions: Other: Biobanking blood; Other: Bone marrow specimens

INTERVENTIONS:
Other: Biobanking blood — Additional volume of 30mL (EDTA) At Screening, pre-Cycle 1 Day 1,Day 1 H8, Day 2, Day of post-cycle 1 and post-cycle 6 evaluation.
Other: Bone marrow specimens — Additional volume of 2mL (EDTA)
  * at screening for correlative studies,at Day 7 for smears and for correlative studies.
  * Post-cycle 1 and post-cycle 6 evaluations for correlative studies.
  Optionnal :
  Trephine biopsy at screening and at post-cycle 1 and 6 evaluations (performed at the same time as aspiration)

SUMMARY:
Acute myeloid leukemia (AML) is a malignancy of aging endowed with poor prognosis. The combination of the hypomethylating agent azacitidine (AZA) with the BCL-2 inhibitor venetoclax (VEN) is the first-line treatment of older AML patients but is endowed with substantial resistance. The project leverages functional precision oncology, single-cell studies and mouse experiments to dissect the mechanisms of primary and adaptive resistance to AZA/VEN. The primary objective is to prospectively validate an ex vivo drug sensitivity testing (DST) assay as predictor of primary resistance to first-line AZA/VEN in 100 unfit AML patients. The study will also explore whether newer DST assays with enhanced niche mimicry can improve on the standard assay.

By serially interrogating the short-term fate of both leukemic and immune cells upon AZA/VEN exposure in patients primed towards refractoriness, transient or prolonged remission, the aim is to dissect the cell-intrinsic and immune-mediated mechanisms of primary versus adaptive resistance. A parallel flow cytometry study will interrogate the role of senescence in AZA/VEN activity. These translational studies will be mirrored by experiments in a transplantable AML model derived from syngeneic mice harboring the age-related Tet2-/- leukemia-predisposing genotype. Lineage tracing single-cell experiments will backtrack AZA/VEN resistance to determine whether it is driven by selection or adaptation. The actionable stress sensor Pml will be invalidated in the same model to determine whether Pml-driven senescence contributes to AZA/VEN anti-leukemic activity in vivo. The project will pave the way to the clinical implementation of functional precision oncology in a high-risk malignancy. By simultaneously interrogating cell-intrinsic and immune-mediated drug resistance in vivo in a prospective patient cohort mirrored by controlled mice experiments, the project will provide a framework for the integrative analysis of drug resistance in cancers.

ELIGIBILITY:
Inclusion Criteria:

* be ≥18 years old,
* have a newly diagnosed AML according to ICC 2022 criteria,

  * patients with AML related to prior chemotherapy or radiotherapy for another cancer will be eligible,
  * patients with MDS/AML per ICC 2022 criteria will be eligible,
* have signed the informed consent form of the eTHEMA observatory trial
* have ≥10% blasts on the bone marrow smear at screening,
* have not received any treatment for AML except for hydroxyurea and/or steroids,

  * Patients having previously received hypomethylating agents for an antecedent myelodysplastic syndrome are ineligible,
* be eligible to AZA/VEN or AZA/IVO therapy, due to general health status,
* have an ECOG performance status ≤ 2,
* be planned to receive azacitidine and venetoclax (AZA/VEN) or azacitidine and ivosidenib (AZA/IVO) as frontline therapy,
* weigh ≥ 40 kg (compliance to Loi Jardé for PB sampling),
* have provided written informed consent obtained prior to any screening procedures

Exclusion Criteria:

At screening, patients must NOT:

* have suspected or proven acute promyelocytic leukemia based on morphology, karyotype or molecular assay, including APL with non-PML::RARA rearrangements,
* have suspected or proven AML with t(9;22)(q34.1;q11.2)/BCR::ABL1 based on karyotype or molecular assay,
* have myeloid sarcoma,
* have failed to perform bone marrow aspiration at screening,
* have received previous therapy for AML with any investigational agent or cytotoxic drug, within 28 days before starting treatment. Only hydroxyurea is permitted for the control of blood counts. Aside from hypomethylating agents, other treatments for an antecedent myeloid neoplasm (MDS or MPN) are not considered as exclusion criteria,
* be pregnant or breastfeeding (for women),
* present any of concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study,
* be enrolled in a clinical trial which could compromise participation in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already included in eTHEMA observationnal cohort
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-06-19 (Estimated); Study Completion 2027-06-19 (Estimated)

PRIMARY OUTCOMES:
Overall Response (CR+CRh+Cri) | Up to 6 months
  Overall Response (CR+CRh+Cri) per European LeukemiaNet 2022 criteria (Döhner et al., Blood 2022), according to DST on the NEXT platform on the population treated per protocol (AZA/VEN).

SECONDARY OUTCOMES:
Number of MRD-negative response (including CRMRD-, CRhMRD- and CRiMRD-) | Up to 6 months
Best response after any number of AZA/VEN cycles | Up to 6 months
  It is ranked as follow : CR > CRh > Cri
MRD-negative response after any number of AZA/VEN cycles | Up to 6 months
  including CRMRD-, CRhMRD- and CriMRD-
Response duration | Up to 6 months
  Defined as the interval between first response among CR, CRh and Cri
Treatment failure per ELN22 criteria | Up to 6 months
Overall survival | Up to 6 months
Event-free survival | Up to 6 months
Relapse-free survival | Up to 6 months
Cumulative Incidence of Relapse (CIR) according to DST on the NEXT platform | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided